CLINICAL TRIAL: NCT02476162
Title: Feasibility of Assessing Blood Pressure Remotely in Childhood Cancer Survivors (Pilot Study-Survivor)
Brief Title: Assessing Blood Pressure Remotely in Childhood Cancer Survivors
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FABRIC; NCI-2015-02265 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-06-16; First posted 2015-06-19 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Hypertension
Keywords: Childhood Cancer Survivor; Cancer Prevention and Control; Blood Pressure Monitoring; Pre-Hypertension
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Daily for 3 Months: Participants randomly assigned to this group will be instructed to measure their blood pressure (BP) every day during the 3-month study period. BP reading will be taken using an iHealth Wireless Blood Pressure Monitor.
  Interventions: Device: iHealth Wireless Blood Pressure Monitor
- Group 2: Daily for 1 Week/Month: Participants randomly assigned to this group will be instructed to measure their BP for seven consecutive days once each month during the 3-month study period. BP reading will be taken using an iHealth Wireless Blood Pressure Monitor.
  Interventions: Device: iHealth Wireless Blood Pressure Monitor
- Group 3: 3 Consecutive Days Once/Month: Participants randomly assigned to this group will be instructed to measure their BP for seven consecutive days once each month during the 3-month study period. BP reading will be taken using an iHealth Wireless Blood Pressure Monitor.
  Interventions: Device: iHealth Wireless Blood Pressure Monitor

INTERVENTIONS:
Device: iHealth Wireless Blood Pressure Monitor — Participants will be provided with an iHealth Wireless Blood Pressure (BP) Monitor and instructions for proper use (based on a standard protocol). The iHealth device pairs easily with a cell phone or other mobile device equipped with the iHealth app (freely available on app stores for both Apple and Android devices). Participants place the cuff on their arm and press start on their mobile device. The device measures BP using the oscillometric method and automatically downloads measurements and timing to a cloud-based server.
  Participants will be educated that individual BP readings can be highly variable and that any one high or low reading has little or no significance. They will also be encouraged not to measure their blood pressure more than twice in the morning and twice in the evening.
  Other Names: Blood Pressure Cuff

SUMMARY:
Second malignant neoplasms and cardiac late effects are primary drivers of serious non-recurrence morbidity and mortality in long term childhood cancer survivors. Cardiac late effects have been most prominently associated with exposure to high doses of anthracyclines or chest radiation. While increased recognition of late effects has resulted in risk-targeted therapy and reductions in use of high dose radiation and anthracyclines for many patients, these cardiotoxic exposures continue to be essential components of curative childhood cancer therapy. In addition, as survivors age they are increasingly susceptible to other general risk factors for cardiovascular disease recognized in the general population, such as hypertension, obesity, dyslipidemia, and diabetes.

This study will evaluate a high blood pressure monitor (HBPM)-based intervention for the early detection of pre-hypertension and prevention of clinical hypertension in survivors of childhood cancer. Eligible and consenting participants will be randomized into one of three groups:

GROUP 1: Instructed to measure blood pressure (BP) every day for 3 months. GROUP 2: Instructed to measure BP for 7 consecutive days once a month, for 3 months.

GROUP 3: Instructed to measure blood pressure for 3 consecutive days each month, for 3 months.

The randomization to the above groups will be done using sequential assignment of newly recruited participants based on a randomly ordered list.

PRIMARY OBJECTIVE:

* Evaluate the feasibility of High Blood Pressure Monitoring (HBPM) for three consecutive months using a remote blood pressure device provided to participants of the St. Jude Lifetime cohort (SJLIFE) protocol.

SECONDARY OBJECTIVES:

* Assess compliance with use of HBPM by measurement frequency, evaluating overall and defined minimum use in each of the three different groups.
* Assess compliance with use of HBPM by cell phone status, evaluating those with and without a personal cell phone capable of connecting directly to the home blood pressure monitoring device via Wi-Fi or Bluetooth network.

DETAILED DESCRIPTION:
The proposed research and testing being done during this study includes:

1. Screening evaluation and consent - Individuals will be asked questions to help the investigators determine if they are eligible to participate. This includes questions about medical history pertaining to blood pressure, medicines, and certain medical conditions, and if the individuals are willing to use the technology provided by the study. For individuals who are eligible to participate, an opportunity will be provided to discuss the study and complete the consent process.
2. Group assignment and randomization - Participants will be randomly assigned to one of three groups: a study team member will select one of sixty identical envelopes, each containing a group assignment, with 20 envelopes containing each of the three group assignments. This random group assignment determines the frequency with which participants will monitor their blood pressure at home. The randomization between three different groups will help investigators determine how often survivors can consistently monitor their blood pressure.
3. Educational session - After participants have been assigned to a group, they will be instructed on how to set up and use the home blood pressure monitoring device.
4. Monitoring blood pressure at home - Participants will be asked to monitor their blood pressure at home in the morning and evening using a remote monitoring device over a three-month period. Frequency of monitoring depends on the random group assignment. The device is the iHealth Wireless Blood Pressure Monitor which is a wireless blood pressure monitoring device that fits snugly around one arm and automatically measures and records blood pressure in about one minute. The device will be paired with the participant's smart phone or study-provided iPod Touch, which is then used to operate the device and save the blood pressure readings. After completion of the three-month monitoring period, participants will be asked to return the device (and iPod Touch, if applicable).
5. Reminders to use the device - Participants are to start monitoring their blood pressure when they return home after completion of their St. Jude visit. During the educational session, participants will be asked to set up reminders on their smart phone or study-provided iPod Touch to alert them to monitor their blood pressure. Depending on how often they are assigned to monitor their blood pressure, they may also receive email and/or text reminders to prompt them to monitor their blood pressure. In addition, a study team member may contact them if they have three or more measurements above 140/90 mm Hg, as that reading is considered hypertensive. A study team member may contact participants if they are not monitoring as specified by their group assignment to attempt to troubleshoot any barriers and/or technical issues.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on the St. Jude protocol: SJLIFE
* Arm circumference between 22-47 cm
* Willing to use and return the technology provided by the study

Exclusion Criteria:

* Medical history of atrial fibrillation or arrhythmia
* Currently taking anti-hypertensive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients at St. Jude Children's Research Hospital who are currently enrolled on the SJLIFE protocol, and who meet all eligibility requirements.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who meet or exceed defined minimum use of HBPM device by group | From Day 0 through 3 months
  The proportion of participants who meet or exceed the defined minimum level of compliance with recording of scheduled blood pressure measurements will be reported. Minimum use is defined as:
  Groups 1 and 2: Successful recording of 12 measurements (maximum 2 per day, one morning and one evening) over any 7 day period in at least 2 of the 3 months of the study.
  Group 3: Successful recording of two measurements each day (morning and evening) for three consecutive days, at least once in each of the 3 months of the study.

SECONDARY OUTCOMES:
Compliance rate for the use of the HBPM device by group measurement frequency | From Day 0 through 3 months
  The overall compliance rate for each group will be calculated as the number of measurements recorded divided by the number of measurements scheduled.
Proportion of participants who comply with the use of HBPM device by cell phone status | From Day 0 through 3 months
  Calculations will be done for participants who own a smart phone compatible with the HBPM device compared to those who need to be supplied with an additional device to pair with the HBPM device. The overall compliance for each group will be calculated as the number of measurements recorded divided by the number of measurements scheduled.
Number of participants who fail to record any blood pressure measurements over the course of a month | From Day 0 through 3 months
Proportion of participants by group who recorded at least 80% of scheduled measurements | From Day 0 through 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Todd M. Gibson, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols